CLINICAL TRIAL: NCT00583804
Title: Implanted Myoelectric Control for Restoration of Hand Function in Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Case Western Reserve University (Other); VA Office of Research and Development (U.S. Federal Agency); FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kevin Kilgore, Program Manager, MetroHealth Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB89-00027; VA Merit Review A3707R (Other Grant/Funding Number: Dept. Veterans Affairs)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury; Tetraplegia
Keywords: Spinal Cord Injury; Tetraplegia; Functional Electrical Stimulation; Neuroprosthesis
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation ON (Experimental): Individuals implanted with stimulator/sensor device. Stimulator is turned on and is active.
  Interventions: Device: IST-12
- Stimulation OFF (Active Comparator): Function with stimulation turned off.
  Interventions: Device: IST-12

INTERVENTIONS:
Device: IST-12 — Implanted stimulator and sensor device, with twelve implanted stimulating electrodes and two myoelectric signal recording electrodes.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an implanted stimulator and sensor for providing hand and arm function for individuals with cervical level spinal cord injury.

DETAILED DESCRIPTION:
The design of this study is to determine the efficacy of improving upper extremity function in tetraplegic subjects after receiving an implantable device for neuromuscular control. Evaluations will be made so as to document changes in performance of manipulative tasks when using the stimulation system.

Subjects who consent to participate in this project will have an implantable stimulator surgically placed in the upper extremity for control of the upper extremity. A series of tests will be performed before implantation, and repeated at intervals after implantation to assess changes in each subject's performance.

This study is a non-randomized feasibility study with concurrent (neuroprosthesis on and off) and longitudinal (pre- and post-implantation/training) self-controls.

Subjects participating in the study can expect to be actively involved in the study for two years after implantation and followed for life thereafter. The screening procedures take up to two days, depending on the specific evaluations necessary to determine candidacy. Pre-surgical exercise is conducted for at least two weeks. The implantation surgery itself lasts one day, with three to seven days of post-surgical hospitalization. Following an eight-week exercise program and a twelve-week training program, subjects are discharged from the active rehabilitation phase. They are followed quarterly for one year, and then annually thereafter.

The device is referred to as the Implanted Stimulator-Telemeter (IST) -12. The device uses functional electrical stimulation (FES) to activate paralyzed muscles.

ELIGIBILITY:
Inclusion Criteria:

* C5-C8 spinal cord injury
* Minimum of one-year post injury with no additional function prior to implantation surgery
* Male or female
* 18-60 years of age
* intact vision
* pharmacologically controlled spasticity, when applicable
* Functional in wheelchair with adequate trunk support to allow bimanual manipulation
* Positive attitude and motivation with supportive home environment
* Willingness to return to laboratory for periodic evaluation and testing
* Free of contractures known to diminish performance of the system (e.g., supination contracture of the wrist).
* Integrity of the lower motor neuron (peripheral nerve) to the muscles to be activated
* Adequate range of motion of joints of the shoulder, wrist, and hand (upper extremity).
* If an acute infection is present, the subject will not be considered for surgery until it clears.

Exclusion Criteria:

* Prior history of a major chronic systemic infection or other illness that would increase the risk of surgery.
* Contraindications include immunologic diseases, cardiac arrhythmias, undiagnosed or high-risk breast masses, dermatologic conditions, and any major system failure.
* Acute infection currently present that has not cleared.
* Hypersensitivity that inhibits their ability to sustain pressure over their digits.
* Blind
* Uncontrolled disorders, i.e., seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1989-04-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2027-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Kilgore, Ph.D., Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Peckham PH, Kilgore KL, Keith MW, Bryden AM, Bhadra N, Montague FW. An advanced neuroprosthesis for restoration of hand and upper arm control using an implantable controller. J Hand Surg Am. 2002 Mar;27(2):265-76. doi: 10.1053/jhsu.2002.30919. PMID 11901386
- [Background] Kilgore KL, Bryden A, Keith MW, Hoyen HA, Hart RL, Nemunaitis GA, Peckham PH. Evolution of Neuroprosthetic Approaches to Restoration of Upper Extremity Function in Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2018 Summer;24(3):252-264. doi: 10.1310/sci2403-252. PMID 29997428
- [Result] Peckham PH, Keith MW, Kilgore KL, Grill JH, Wuolle KS, Thrope GB, Gorman P, Hobby J, Mulcahey MJ, Carroll S, Hentz VR, Wiegner A; Implantable Neuroprosthesis Research Group. Efficacy of an implanted neuroprosthesis for restoring hand grasp in tetraplegia: a multicenter study. Arch Phys Med Rehabil. 2001 Oct;82(10):1380-8. doi: 10.1053/apmr.2001.25910. PMID 11588741
- [Result] Kilgore KL, Hoyen HA, Bryden AM, Hart RL, Keith MW, Peckham PH. An implanted upper-extremity neuroprosthesis using myoelectric control. J Hand Surg Am. 2008 Apr;33(4):539-50. doi: 10.1016/j.jhsa.2008.01.007. PMID 18406958
- See also: Cleveland FES Center — http://fescenter.org/index.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Implanted Individuals: Individuals implanted with stimulator/sensor device. These individuals were implanted with the IST-12 device. The IST-12 is an implanted stimulator and sensor device, with twelve implanted stimulating electrodes and two myoelectric signal recording electrodes. The device was implanted in the chest, hand and arm to provide functional grasp and reach.
  All participants received the implanted device. During the primary outcome testing, the device was tested with the device "on" and active and compared with the results when the device was turned off. No blinding of either the subject or evaluator was possible because of the obvious response when the stimulator is on (i.e. the hand opens and closes when the stimulator is on; the hand is paralyzed when the stimulator is off).
Period: Overall Study
Arm/Group | Implanted Individuals
Started | 10
Completed | 10 (Subjects were considered enrolled when they underwent implantation of the device. All completed.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Implanted Individuals: Individuals implanted with stimulator/sensor device.
  IST-12: Implanted stimulator and sensor device, with twelve implanted stimulating electrodes and two myoelectric signal recording electrodes.
Arm/Group | Implanted Individuals
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 37 [26 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Grasp-Release Test - Baseline [Median (Full Range); unit: Objects] — The Grasp-Release tests consists of six standard objects requiring different grasp patterns and forces to pick up and move. The subjects have a fixed period of time to attempt to acquire the object and move it from one location on the test board to a second location. The outcome is measured as the number of objects that they can successfully pick up and move. The minimum score is 0 and the maximum score is 6.
  Objects | 2 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Grasp-Release Test
Description: Grasp and Release Test (GRT) - The Grasp and Release Test (GRT) [Wuolle, 1994; Smith et al., 1996; Carroll et al., 2000; Taylor et al., 2002; Mulcahey et al., 2004], developed at the Cleveland FES Center, has been utilized by multiple centers to show improvements in hand function after implantation of a neuroprosthesis and tendon transfers [Peckham, 2001]. This pick-and-place test requires the participant to unilaterally acquire, move, and release six objects varying in weight and size. The objects are: 1) a small peg, 2) a wooden cube, 3) a small juice can, 4) a videotape, 5) a paperweight (~1000g) and a simulated fork task (spring-loaded plunger). The number of objects that the participant can successfully manipulate are scored. Success in manipulating each object in the GRT is defined as the ability to pick up and place the object at least once within 30 seconds.
Time Frame: One Year
Measure: Median (Full Range); unit: Number of Objects
Arm/Group | Stimulation ON | Stimulation OFF
Number analyzed (Participants) | 10 | 10
Number of Objects | 5.5 [5 to 6] | 2 [0 to 4]

2. Primary Outcome: Activities of Daily Living Test
Description: The ADL Abilities Test was developed to measure differences in activity performance with and without a hand neuroprosthesis. Scoring is based on an activity analysis approach. The activities, which are chosen by the participant, are broken down into phases, and each phase is scored for the amount of assistance the participant uses: 1) "Physical Assistance" (PA): assistance from an attendant, 2) "Adaptive Equipment" (AE): any modifications of the activity or its components, 3) "Orthotic Assistance" (OA): an orthotic device that the participant normally wears all day (e.g., a dorsal wrist support), and that can be considered a modification of the hand, 4) "Self Assistance" (SA): use of any part of the body other than the dominant hand, or use of the test equipment in an adapted way to complete the activity (e.g., using two hands to hold a glass, or sliding an object to the end of the table for grasping), and 5) "Independent".
Time Frame: Three months
Measure: Median (Full Range); unit: Number of Tasks Improved
Groups:
- Implanted Individuals: Individuals implanted with stimulator/sensor device. These individuals were implanted with the IST-12 device. The IST-12 is an implanted stimulator and sensor device, with twelve implanted stimulating electrodes and two myoelectric signal recording electrodes. The device was implanted in the chest, hand and arm to provide functional grasp and reach.
Arm/Group | Implanted Individuals
Number analyzed (Participants) | 10
Number of Tasks Improved | 6 [2 to 11]

3. Secondary Outcome: Adverse Events
Description: Self-reported adverse events.
Time Frame: From date of implant until study completion or date of death from any cause.
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Implanted Individuals: Individuals implanted with stimulator/sensor device.
  IST-12: Implanted stimulator and sensor device, with twelve implanted stimulating electrodes and two myoelectric signal recording electrodes.
  Note that all subjects received the implanted device and used the device in the laboratory and at home throughout the course of the study. Therefore there is only a single Arm for adverse events - all subjects received the intervention and stimulation.
Arm/Group | Implanted Individuals
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Individuals (N=10)
Device infection (Infections and infestations) | 2 (2) — Device infection requiring removal of some or all of implanted components.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes